CLINICAL TRIAL: NCT00377104
Title: A Phase I Dose-Escalation Study of Flavopiridol (NSC 649890) Administered as a 30 Minute Loading Dose Followed by a 4-Hour Infusion in Patients With B-Cell Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) Following Cytoreduction With Chemotherapy
Brief Title: Alvocidib in Treating Patients With B-Cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00161; OSU 05116; OSU-IRB-2006C0031; CDR0000501975; OSU-05116; U01CA076576 (NIH); NCT01645579 (obsolete NCT alias)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Contiguous Stage II Small Lymphocytic Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — alvocidib

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive alvocidib IV over 30 minutes (loading dose), followed by alvocidib IV over 4 hours on days 1, 8, and 15. Treatment repeats every 5 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of flavopiridol in treating patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma. Drugs used in chemotherapy, such as alvocidib, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity profile, dose-limiting toxicity, and maximum tolerated dose of flavopiridol (alvocidib) as consolidation chemotherapy after cytoreduction chemotherapy in patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics and cellular pharmacodynamics of flavopiridol in these patients.

II. Determine the complete response (CR) and overall response rate (CR and partial response) of patients treated with flavopiridol.

OUTLINE: This is a dose-escalation study. Patients receive alvocidib intravenously (IV) over 30 minutes (loading dose), followed by alvocidib IV over 4 hours on days 1, 8, and 15.

Treatment repeats every 5 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 12 patients are treated at the MTD (i.e., recommended phase II dose). Patients undergo blood collection at baseline and periodically during study for pharmacokinetic and cytokine studies (levels of tumor necrosis factor-alpha, interleukin [IL]-6, -11, and -16) by enzyme-linked immunosorbent assay (ELISA). Interphase cytogenetics, p53 mutational status, p53/ATM function, V_H mutational status, zeta-chain-associated protein kinase 70 (ZAP-70) overexpression, and single nucleotide polymorphisms are also examined.

After completion of study treatment, patients are followed at 2 months and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * B-cell chronic lymphocytic leukemia (CLL)
  * Small lymphocytic lymphoma (SLL)
* Must have received 1-3 prior therapies for CLL

  * Completed therapy 2-12 months ago
  * Prior therapy must have led to a partial response or greater
  * No evidence of progressive disease
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm³
* WBC ≤ 5,000/mm³
* Platelet count ≥ 50,000/mm³
* Cytopenia allowed
* Creatinine < 2.0 mg/dL
* Bilirubin ≤ 1.5 times normal (unless due to Gilbert's disease or hemolysis)
* AST ≤ 2 times normal (unless due to hemolysis)
* No secondary malignancy or other disease that would limit survival to < 2 years
* No history of inflammatory bowel disease unless inactive for > 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* No other concurrent chemotherapy
* No concurrent radiotherapy
* No concurrent dexamethasone or other corticosteroid-based antiemetics
* No concurrent chronic corticosteroid therapy
* No other concurrent hormonal therapy except for the following:

  * Steroids for new adrenal failure
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Toxicity profile of alvocidib administered as a 30 minute loading dose followed by a 4-hour infusion once weekly for 3 consecutive weeks every 5 weeks as consolidation therapy following cytoreduction chemotherapy | Day 1, every 2 courses, at 2 months and then every 3 months for 5 years after completion of study treatment
  Assessed utilizing the NCI Common Terminology Criteria for Adverse Events version 3.0.
Dose-limiting toxicity of alvocidib as consolidation chemotherapy after cytoreduction chemotherapy in patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma | Course 1
  The National Cancer Institute Common Toxicity Criteria version 3.0 will be used to characterize toxicity. If no patients experience dose-limiting toxicity, dose escalation will occur. If 1 patient has a dose limiting toxicity, 3 additional patients will be enrolled at that dose. If fewer than 2 of 6 patients experiences dose limiting toxicity, then the next highest dose level will be used for the subsequent cohort of 3 patients. If at any dose level two or more of the six patients experience a dose limiting toxicity, 3 additional patients will be treated at the previous dose level.

SECONDARY OUTCOMES:
Pharmacokinetics and cellular pharmacodynamics of alvocidib administered in this schedule | Baseline and day 1
  Cytokine studies will be examined by standard ELISA assays to determine if increase IL-6 correlates with hypotension, hypoxemia, and tachycardia observed following treatment and to identify the source of production of this cytokine. We will examine interphase cytogenetics, p53 mutational status, p53/ATM functional assay, VH mutational status, and ZAP-70 over-expression.
Complete response (CR) and overall response rate (CR and partial response) of alvocidib in patients with previously-treated CLL | Baseline, every 2 courses, at 2 months and then every 3 months for 5 years after completion of study treatment
  Criteria for response will utilize the Revised National Cancer Institute-sponsored Working Group Guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Andritsos, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Awan FT, Jones JA, Maddocks K, Poi M, Grever MR, Johnson A, Byrd JC, Andritsos LA. A phase 1 clinical trial of flavopiridol consolidation in chronic lymphocytic leukemia patients following chemoimmunotherapy. Ann Hematol. 2016 Jun;95(7):1137-43. doi: 10.1007/s00277-016-2683-1. Epub 2016 Apr 27. PMID 27118540